CLINICAL TRIAL: NCT04895319
Title: Adherence to Computer-assisted Surgical Planning in 136 Maxillofacial Reconstructions
Brief Title: Adherence to Computer-assisted Maxillofacial Reconstructions
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Hongyang Ma, Principle investigator, KU Leuven
Other Study IDs: S63615-3
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Maxillofacial Abnormalities; Computer-assisted Surgery; Virtual Surgical Planning
Keywords: Computer-Assisted Surgery; Treatment Adherence and Compliance; Patient-Specific Modelling
MeSH Terms: conditions — Maxillofacial Abnormalities; Treatment Adherence and Compliance | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Computer-assisted surgery — The reconstruction was performed with the help of virtual surgical plan and 3D printed models.

SUMMARY:
The study was approved by the Local Ethics Committee and was conducted in compliance with the World Medical Association Declaration of Helsinki on medical research. A total of 335 patients who underwent oral and maxillofacial reconstruction were recorded from Jan 2014 to Jun 2020. Reconstruction with computer-assisted surgery ( CAS), which included, virtual surgical planning, computer-aided design-computer-aided manufacturing (CAD-CAM) surgical guides/templates and pre-bent plates on 3D printed models. Reasons for tissue defect were oncologic, osteoradionecrosis, trauma and osteoporosis. Patients undergoing dental implant placement and orthognathic surgery were excluded. Finally, 136 patients were selected and the reasons for partial or abandon surgical plan performance were described and analyzed.

DETAILED DESCRIPTION:
computer-aided design

ELIGIBILITY:
Inclusion Criteria:

1. Maxillofacial reconstruction with CAS, including virtual surgical planning, CAD-CAM surgical guides/templates and pre-bent plates on 3D printed models.
2. Reasons for reconstruction were oncologic, osteoradionecrosis, trauma and osteoporosis.

Exclusion Criteria:

1. Patients undergoing computer-assisted implant surgery were excluded.
2. Patients undergoing computer-assisted orthognathic surgery were excluded.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 136 patients who undergone computer-assisted maxillofacial reconstructive surgeries that conducted from June 2014 to June 2020.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
The adherence of computer-assisted surgery | The outcome were recorded preoperatively or intraoperatively
  The original plans were classified as completely executed, partially executed or abandoned.